CLINICAL TRIAL: NCT00723723
Title: Compliance With LDL-Lowering Therapy For Secondary Prevention of Coronary Heart Disease in Real Life Practice
Brief Title: Compliance With LDL-Lowering Therapy (Study P05467)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05467
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Coronary Heart Disease; Hypercholesterolemia; Hyperlipidemia
MeSH Terms: conditions — Coronary Disease; Hypercholesterolemia; Hyperlipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with coronary heart disease: Patients being treated with a statin for secondary prevention of coronary heart disease
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Statin

SUMMARY:
This observational study is being conducted in patients receiving statin treatment as secondary prevention of coronary heart disease under the current standard of care in compliance with European guidelines. The purpose of the study is to evaluate the percentage of these patients that reach target LDL levels. Additionally this study will measure the patient's compliance to treatment as assessed by counting the returned tablets. Both assessments will be made at visits conducted 6-8 weeks after the first visit and 28-32 weeks after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* 18 years of age or more
* clinically established cardiovascular disease to be considered as patients in secondary prevention
* prior therapy with any statin without achieving goal (2.5 mmol/L of LDL cholesterol) at last lipid check performed

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with a statin for secondary prevention of coronary heart disease
Sampling Method: Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
percentage of patients reaching target LDL levels | 6-8 weeks after first visit and 28-32 weeks after first visit

SECONDARY OUTCOMES:
measure patient compliance to treatment as assessed by counting returned tablets | 6-8 weeks after first visit and 28-32 weeks after first visit